CLINICAL TRIAL: NCT03343080
Title: Lidocaine as an ETT Cuff Media in the Immediate Post-operative Cardiac Surgery Patient Population, and Its Effect on Sedation/Analgesia Requirements: a Pilot Study
Brief Title: Lidocaine as an Endotracheal Tube (ETT) Cuff Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Troy G. Seelhammer, Assistant Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-000621
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Disease
Keywords: Cardiac Surgery
MeSH Terms: conditions — Heart Diseases | interventions — Lidocaine; Sodium Bicarbonate; Air

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buffered Lidocaine (Experimental): At the induction of anesthesia, patients will be breathing 100% oxygen via a face mask and then, become anesthetized according to a standard protocol and at the discretion of the attending anesthesiologist.
  For cardiac surgery patients randomized to the buffered lidocaine arm, the operating room registered respiratory therapist (OR RRT) will inflate the endotracheal tube cuffs with the study drug containing 1.8% lidocaine plus 0.76% sodium bicarbonate until abatement of the air leak at 20 cm of water.
  The intervention will take place while in the operating room. The room nurse anesthetist (CRNA) or anesthesiologist will be aware of the amount of solution instilled in the ETT cuff. The patient will remain intubated after the surgery is complete and will be taken to the cardiac surgical ICU.
  Interventions: Drug: 1.8% lidocaine plus 0.76% sodium bicarbonate
- Air (Placebo Comparator): At the induction of anesthesia, patients will be breathing 100% oxygen via a face mask and then, become anesthetized according to a standard protocol and at the discretion of the attending anesthesiologist.
  For cardiac surgery patients randomized to the air arm, the operating room registered respiratory therapist (OR RRT) will inflate the endotracheal tube cuffs with air until abatement of the air leak at 20 cm of water.
  The intervention will take place while in the operating room. The room nurse anesthetist (CRNA) or anesthesiologist will be aware of the amount of air in the ETT cuff. The patient will remain intubated after the surgery is complete and will be taken to the cardiac surgical ICU.
  Interventions: Other: Air

INTERVENTIONS:
Drug: 1.8% lidocaine plus 0.76% sodium bicarbonate — At the time of intubation, the endotracheal tube cuff will be inflated with a solution containing 1.8% lidocaine plus 0.76% sodium bicarbonate until loss of air leak at a positive pressure of 20 cm of water. This solution will remain in situ through the duration of cardiac surgery, transportation to the intensive care unit, and continued to the time of extubation.
  Arms: Buffered Lidocaine
Other: Air — At the time of intubation, the endotracheal tube cuff will be inflated with air until loss of air leak at a positive pressure of 20 cm of water. The air will remain in situ through the duration of cardiac surgery, transportation to the intensive care unit, and continued to the time of extubation.
  Arms: Air

SUMMARY:
Researchers will compare the effects of lidocaine versus air, as a way to fill the breathing tube cuff which is gently inflated to hold in place the trachea (airway) during surgery. Air is the traditional method used to inflate the breathing tube cuff. Researchers wish to find if lidocaine works better than air to facilitate tolerance to the breathing tube (decreased coughing, sore throat, hoarseness). They also want to learn more about its effectiveness for this particular surgical intervention.

DETAILED DESCRIPTION:
At the induction of anesthesia, Participants will be breathing 100% oxygen via a face mask and then, become anesthetized according to a standard protocol and at the discretion of the attending anesthesiologist. Participants will be receive fentanyl, lidocaine and either succinylcholine or vecuronium to facilitate tracheal intubation. Laryngoscopy will then be performed and the trachea intubated with a standard cuffed ETT. Inflation of the ETT cuff will be performed in accordance with the randomization of either air or 1.8% lidocaine/0.76% solution until such time as there is no air leak around the tube when administering positive pressure to 20 cm H2O. Anesthesia will be maintained with volatile anesthetic with or without a Propofol infusion. Vecuronium will be used to maintain the ulnar nerve train-of-four at 0-3 of four twitches. Lungs will be mechanically ventilated with tidal volumes of 6-8 mL/kg to maintain end-tidalCO2 concentration at 30-35 mm Hg. Anesthesia maintenance will occur until the near end of the surgical procedure. The volatile anesthetic will be discontinued and Propofol will be initiated via a continuous infusion to facilitate transportation to the intensive care unit (ICU). After arrival to the ICU, Neuromuscular blockade will then be antagonized with neostigmine and glycopyrrolate, and the pharynx being gently suctioned under direct vision. Mechanical ventilation to be maintained until swallowing or spontaneous respiration begins, and then, converted to assisted manual ventilation. Extubation will be performed when all of the following criteria are met: 1) full reversal of neuromuscular block (ulnar nerve T4/T1 ratio 1:1, with sustained tetanus at 50 Hz for 5 s and no fade); 2) spontaneous ventilation; and 3) the ability to follow verbal commands (eye opening or hand grip) or demonstrate purposeful unilateral movement (attempting self-extubation); 4) demonstration of hemodynamic stability; 5) adequate hemostasis with combined chest tube output < 100 ml/hour.

The Participant then will be closely monitored as a 1:1 by the room nurse, and by other staff (respiratory therapist, and ICU fellows and consultants) for toleration of the ventilator (coughing, double triggering, "bucking," etc.). on the cardiac surgical intensive care unit. Sedation amount will be recorded electronically once the patient lands in the ICU, until the time of extubation. A member from the study team will physically record "yes," or "no," on the form provided regarding the patient coughing, complaining of a sore throat or difficulty swallowing, having hoarseness or difficulty speaking.

ELIGIBILITY:
Patients who meet the inclusion criteria below and are expected to require ventilatory support for a period of less than 5 hours post-operatively in the cardiac ICU will be enrolled.

Inclusion Criteria:

* All patients > 18 years of age (male and female) who will receive general anesthesia for cardiac surgery at St. Mary's Hospital (SMH) in Rochester, Minnesota
* Cardiac surgery includes: single valve repair, myectomy, cabbage, pericardectomy.
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Age < 18 years old at time of surgery
* Patients who are not sent to the cardiac ICU post-operatively
* Patients who are anticipated to have a difficult tracheal intubation
* Patients having risk factors of postoperative aspiration of gastric contents
* Patients who have respiratory disease or recent respiratory tract infection
* > 1 attempt to secure an airway
* Patients undergoing transcatheter aortic valve replacement (TAVR) procedures or any form of "robotic" procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Troy G Seelhammer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered Lidocaine: 1.8% lidocaine plus 0.76% sodium bicarbonate: At the time of intubation, the endotracheal tube cuff will be inflated with a solution containing 1.8% lidocaine plus 0.76% sodium bicarbonate until loss of air leak at a positive pressure of 20 cm of water
- Air Only: Air: At the time of intubation, the endotracheal tube cuff will be inflated with air until loss of air leak at a positive pressure of 20 cm of water. The air will remain in situ through the duration of cardiac surgery, transportation to the intensive care unit, and continued to the time of extubation.
Period: Overall Study
Arm/Group | Buffered Lidocaine | Air Only
Started | 14 | 18
Completed | 14 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buffered Lidocaine | Air Only | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (14.9) | 59.4 (16.6) | 60.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Total Sedation Requirements
Description: Total amount of Propofol dose used as measured in total milligrams.
Time Frame: baseline through extubation
Population: Only 10 subjects in the buffered lidocaine arm and 13 subjects in the air only arm received Propofol for sedation. The remaining subjects received other sedation drugs per physician discretion.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Buffered Lidocaine | Air Only
Number analyzed (Participants) | 10 | 13
milligrams | 325 (248) | 1158 (1426)

2. Secondary Outcome: Total Duration of Mechanical Ventilation
Description: Total amount of time that the participant is intubated as measured in minutes.
Time Frame: baseline through extubation
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Buffered Lidocaine | Air Only
Number analyzed (Participants) | 14 | 18
minutes | 499 [440 to 613] | 529 [380 to 700]
Statistical Analysis 1: Comparison: Buffered Lidocaine vs Air Only; Test type: Superiority; p = 0.776, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Richmond Agitation-Sedation Score (RASS)
Description: The Richmond Agitation-Sedation Scale (RASS) is a medical scale used to measure the agitation or sedation level of a patient.. It is a 10-point scale comprised of four levels of agitation (+1 to +4), one level defining a calm and alert state (0) and five levels of sedation (-1 to -5). The higher the positive number (+) the more agitated or combative a patient is and the higher the negative number (-) the deeper the sedation of the patient.
Time Frame: 4 hours post-extubation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buffered Lidocaine | Air Only
Number analyzed (Participants) | 14 | 18
score on a scale | -0.2 (0.4) | -0.4 (0.5)
Statistical Analysis 1: Comparison: Buffered Lidocaine vs Air Only; 4 hours post-extubation; Test type: Superiority; p = 0.296, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline to 4 hours post extubation for each subject.
Arm/Group | Buffered Lidocaine | Air Only
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 14/14 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buffered Lidocaine (N=14) | Air Only (N=18)
Agitation or restlessness (General disorders) | 0 (0) | 1 (1)
Difficulty swallowing (General disorders) | 1 (1) | 2 (2)
Hoarseness present (General disorders) | 10 (10) | 15 (15)
Cough (General disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT03343080/Prot_SAP_000.pdf